CLINICAL TRIAL: NCT01686880
Title: Treatment With Yttrium90 Radioembolization Prior to Surgical Resection or Radiofrequency for Hepatocellular Carcinoma in Cirrhotic Liver
Brief Title: Y90 Radioembolization Prior to Surgical Resection or Radiofrequency for Hepatocellular Carcinoma in Cirrhotic Liver
Acronym: TRYPHON
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment and an unexpected low treatment rate
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRYPHON
Record Dates: First submitted 2012-09-11; First posted 2012-09-18 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis
Keywords: Hepatocellular Carcinoma; Liver Cirrhosis; radioembolization; SIRT; TARE; Sirspheres; neoadjuvant; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preoperative aTARE (Experimental): The patients in this arm will receive Sirsphere trans-arterial radioembolization before surgery
  Interventions: Device: Sirsphere trans-arterial radioembolization

INTERVENTIONS:
Device: Sirsphere trans-arterial radioembolization — Patients will receive Sirsphere trans-arterial radioembolization before surgery
  Other Names: TARE; SIRT

SUMMARY:
The purpose of this study is to assess the safety of transarterial radioembolization prior to surgical resection or radiofrequency in cirrhotic patients with hepatocellular carcinoma

DETAILED DESCRIPTION:
The purpose of this study is to assess the peri-operative morbidity and mortality of supraselective ablative transarterial radioembolization prior to surgical resection or radiofrequency in cirrhotic patients with HCC

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Cirrhotic liver demonstrated by typical liver dysmorphy on imaging and/or liver biopsy.
* HCC with at least one lesion measuring more than 1 cm in diameter with a single dynamic imaging technique (CT or MRI), showing intense arterial uptake followed by washout of contrast in the venous-delayed phases, or diagnosed by biopsy.
* Borderline resectable disease eligible for surgical resection or radiofrequency destruction.
* No extra-hepatic dissemination.
* ECOG Performance status < 2.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Signed written informed consent (approved by an Independent Ethics Committee) obtained prior to any study specific baseline procedures.

Exclusion Criteria:

* Decompensated cirrhosis (Child Pugh B, C).
* Extra-hepatic tumour spread.
* Previous or concomitant malignancies within five years other than basal cell carcinoma of the skin.
* Pregnancy, lactation or refusal to use adequate contraceptive measures (hormonal or barrier method of birth control, abstinence).
* Pre-existing other hepatic disease (liver abscess, hepatic sarcoidosis or tuberculosis, sclerosing cholangitis, …).
* Previous trans-arterial radioembolization (TARE).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition of the administered materials.
* Bleeding diathesis, history of cardiovascular ischemic disease or cerebrovascular incident within the last six months.
* Major surgery within four weeks.
* Uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Uncontrolled Diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Peri-operative morbidity | 3 months after surgery
  peri-operative morbidity of supraselective ablative transarterial radioembolization prior to surgical resection or radiofrequency in cirrhotic patients with HCC (starting from date of inclusion till 90 days after surgery or hospital discharge if more than 90 days)

SECONDARY OUTCOMES:
Survival | 3 years
  Assessment of the overall disease free survival and Overall Survival
One and three years survival | one and three years
  Estimation of disease free survival and overall survival rates after 1 and 3 years
Tumor regression | 8 weeks after Trans-arterial radioembolization
  Assessment of tumour size regression after Trans-arterial radioembolization by MRI
Functional Imaging | 3 years
  Assessment of imaging parameters changes (DW-MRI, FDG-PET/CT) and MAA-SPECT-CT in relation to the outcome measured by tumour regression after TARE, disease free and overall survival.
Contra-lateral Lobe Hypertrophy | 3 Years
  Assessment of TARE induced liver contralateral lobe hypertrophy (volumetric measurement by MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Alain Hendlisz, MD, Principal Investigator — Jules Bordet Institute; Vincent Donckier, MD, PHD, Principal Investigator — Erasme University Hospital
Locations (2):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Erasme Hosptial, Brussels

REFERENCES:
- [Derived] Lemaire M, Lucidi V, Bouazza F, Katsanos G, Vanderlinden B, Levillain H, Delatte P, Garcia CA, Vouche M, Galdon MG, Demetter P, Deleporte A, Hendlisz A, Flamen P, Donckier V. Selective internal radiation therapy (SIRT) before partial hepatectomy or radiofrequency destruction for treatment of hepatocellular carcinoma in cirrhotic patients: a feasibility and safety pilot study. HPB (Oxford). 2018 Jul;20(7):641-648. doi: 10.1016/j.hpb.2018.01.006. Epub 2018 Feb 24. PMID 29486918
- See also: Jules Bordet Institute — http://www.bordet.be/
- See also: Erasme Hospital — http://www.erasme.ulb.ac.be/